CLINICAL TRIAL: NCT03574298
Title: Effect of Radical Prostatectomy on Involuntary Pelvic Floor Muscle Contraction
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon hospital, Pierre and Marie Curie University
Other Study IDs: P GREEN 0001
Record Dates: First submitted 2018-06-18; First posted 2018-06-29 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Radical prostatectomy; urinary incontinence; pelvic floor muscle; reaction time
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluate the effect of radical prostatectomy on involuntary pelvic floor muscle contraction

DETAILED DESCRIPTION:
Radical prostatectomy may cause stress urinary incontinence (SUI). That poses problem in terms of quality of life. There are many treatment options available for patients with SUI, but the exact mechanism is not known. We compared, in continent and incontinent men post-radical prostatectomy, the correlation between the temporal course of pelvic floor activation during cough.

Simultaneously, recordings of electromyographic activity of external anal sphincter (EAS EMG) and external intercostal muscle (EIC EMG) during coughing will be made with a pair of pre-gelled electrodes. Cough effort cause an involuntary pelvic contraction. Intercostals muscles recording was chosen because they are one of the muscular components of cough initiation with diaphragm muscle. 24h pad-weighing test is used to quantify urinary incontinence. We will measure the latency between the onset of the EIC EMG and the EAS EMG (RT3), during a cough effort. We will also measure the duration of the contraction, the maximum EAS EMG activity and the area under the curve.

ELIGIBILITY:
Inclusion Criteria:

* Follow in neuro-urology for lower urinary tract symptoms
* Radical Prostatectomy

Exclusion Criteria:

* Perineal Radiotherapy
* Surgery for stress urinary incontinence

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting for urodynamic assessment
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Latency (time) | 1 day: During electromyographic recording
  The time (latency) between the onset of the external intercostal muscle (EIC EMG) and the electromyographic activity of external anal sphincter (EAS EMG), during a cough effort.

SECONDARY OUTCOMES:
Duration (time) | 1 day: During electromyographic recording
  The duration of contraction of external anal sphincter (defined as the time between the onset of the electromyographic activity of external anal sphincter and the end of the electromyographic activity of external anal sphincter).
Maximum | 1 day: During electromyographic recording
  The maximum of contraction of the electromyographic activity external anal sphincter.
Area under the curve | 1 day: During electromyographic recording
  the area under the curve of the electromyographic activity external anal sphincter.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — GREEN GRC-01, Neuro-urology, hôpital Tenon
Locations (1):
- Department of Neuro-urology, Tenon hospital, Paris, France